CLINICAL TRIAL: NCT01211704
Title: Paliperidone Palmitate Efficacy and Safety in Bipolar Disorder Complicated by Alcoholism: A Double-blind, Placebo-controlled, Randomized, Parallel Groups, Multi-center Study.
Brief Title: Paliperidone Palmitate Efficacy and Safety in Bipolar Disorder Complicated by Alcoholism
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Miami (Other)
Collaborators: Ortho-McNeil, Inc. (Industry)
Responsible Party: Principal Investigator, Ihsan Salloum, Professor of Psychiatry, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20081123
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Bipolar Disorder
Keywords: Bipolar, Alcoholism
MeSH Terms: conditions — Bipolar Disorder; Alcoholism | interventions — Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo, Counceling (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Paliperidone Palmitate (Experimental): Paliperidone Palmitate
  Interventions: Drug: Paliperidone Palmitate

INTERVENTIONS:
Drug: Paliperidone Palmitate — NVEGA® SUSTENNA™ or placebo in equivalent ml doses according to the following schedule: Day 1: INVEGA® SUSTENNA™ 234mg vs. placebo injection (equivalent ml); Day 8 (week 1) INVEGA® SUSTENNA™ 156mg vs. placebo injection (equivalent ml); Day 36 (week 5): INVEGA® SUSTENNA™ 117 mg vs. placebo injection (equivalent ml) ( this latter dose could range from 39mg to 156mg according to tolerability and clinical symptoms of bipolar disorder). Treatment with INVEGA® SUSTENNA™ /Placebo will last 5 weeks.
  Other Names: INVEGA® SUSTENNA™
  Arms: Paliperidone Palmitate
Drug: Placebo — Placebo in equivalent ml doses to experimental intervention (Paliperidone Palmitate)
  Arms: Placebo, Counceling

SUMMARY:
The primary specific aim is to examine the efficacy of Paliperidone extended release Paliperidone Palmitate Injection (INVEGA® SUSTENNA™) compared to placebo in decreasing manic symptoms in patients with comorbid DSM-IV bipolar disorder and alcohol dependence. The investigators hypothesize that the Paliperidone Palmitate Injection (INVEGA® SUSTENNA™) treated group will have a statistically significant advantage on improvement in manic symptoms. They will also have higher rate of treatment response and remission.

DETAILED DESCRIPTION:
Subjects who meet study inclusion criteria will be randomized to receive an add-on Paliperidone Palmitate ( INVEGA® SUSTENNA™ ) according to the following schedule described in the medication prescribing information: INVEGA® SUSTENNA™ (PALIPERIDONE PALMITATE) Extended-Release Injectable Suspension ). Tolerability of the paliperidone will be established by either 1) a documented history of having taken either paliperidone or risperidone in the past without any untoward effects or allergic reactions, or 2) by prescribing oral paliperidone 6mg per day for three days with absence of any allergic or severe untoward side effects for those with no prior history of having taken these medications, prior to initiating treatment with INVEGA® SUSTENNA™ according to the manufacturers' recommendations.

Eligible patients will be randomized to INVEGA® SUSTENNA™ or placebo in equivalent ml doses according to the following schedule: Day 1: INVEGA® SUSTENNA™ 234mg vs. placebo injection (equivalent ml); Day 8 (week 1) INVEGA® SUSTENNA™ 156mg vs. placebo injection (equivalent ml); Day 36 (week 5): INVEGA® SUSTENNA™ 117 mg vs. placebo injection (equivalent ml) ( this latter dose could range from 39mg to 156mg according to tolerability and clinical symptoms of bipolar disorder); Day 64 (week 9) no injection; weeks 10 and 11 safety assessment follow-up ( see Study Schematics below). Both treatment groups will participate in standardized individual medication adherence counseling. Subjects with bipolar disorder and who are actively drinking will be recruited into the study. Subjects who have been stable on treatment as usual medications for bipolar disorder for at least three weeks, and who meet all the inclusion criteria will be randomized to receive the double blind study medication consistent of either Paliperidone Palmitate injection ( INVEGA® SUSTENNA™ )or placebo (1:1 ratio). To optimize the likelihood of balanced groups, the investigators will use urn randomization with the following variables: Gender (males vs. females), treatment as usual medication (divalproex sodium vs. other mood stabilizers), presenting bipolar subtype (manic vs mixed) and baseline drinking severity (< vs. > 50% heavy drinking days (> 4 standard drinks for females and > 5 standard drinks per males) in the month prior to enrollment). After randomization, subjects will be assessed weekly at weeks 1, 2, 3, 4, 5, 6, 7, 8,9 of the double-blind treatment phase a and at week 10 and 11 for safety observation follow-up.. The investigators propose to test the above hypotheses in 75 subjects at three sites (25 subjects per site) All subjects will receive a weekly Standardized supportive individual medication adherence counseling session.

ELIGIBILITY:
Inclusion Criteria: Patients will be assessed using the Mini International Neuropsychiatric Interview at baseline, which will be carried out at least three days after all acute withdrawal symptoms have cleared. Subjects who meet DSM-IV criteria for alcohol use disorder (abuse or dependence) and a concurrent bipolar I disorder, (Mixed or Mania State) and a score on the YMRS of 16 or above, and without any exclusion criteria will be recruited for the study. The following criteria must be met. A) Abstinent from alcohol not to exceed 21 consecutive days, and a score of <8 on the CIWA-Ar, [Sullivan, 1989 #1412] at the time of randomization. B) An average minimum of > 7 drinks per week for females or > 14 drinks per week for males, over a consecutive 4-week period during the 12-week period prior to baseline. C) A breath alcohol concentration (BAC) of 0 at the time of signing Informed Consent. D) Subject stable on treatment as usual medications for bipolar disorder for at least three weeks prior to randomization.

-

Exclusion Criteria: Patients with the following disorders will be excluded from the study: 1) Schizophrenia, schizoaffective, and any non-bipolar psychotic disorder, unipolar major depression, primary anxiety disorders, mental retardation, and signs of impaired cognitive functioning (operationalized as a score < 25 on Folstein's Mini-Mental Status Exam). [Folstein, 1975 #1179]. 2) Current DSM-IV criteria for dependence on substances other than alcohol, cannabis, nicotine, or caffeine. 3) Neurological conditions including epilepsy, history of brain injury, encephalitis, or any organic brain syndrome or documented focally abnormal electroencephalograph examination (EEG), or recent history (within the past two years) of alcohol withdrawal seizure. 4) Medical conditions including severe cardiac, liver, kidney, endocrine (e.g. diabetes), hematologic (e.g. porphyria or any bleeding abnormalities), or other impairing medical conditions, or impending surgery. 5) Congenital prolongation of the QT interval (congenital long QT syndrome), and a history of cardiac arrhythmias or other conditions that prolong the QT interval such as bradycardia; hypokalemia or hypomagnesemia; or on concomitant medications known to prolong QTc including Class 1A (e.g., quinidine, procainamide) or Class III (e.g., amiodarone, sotalol) antiarrhythmic medications, antipsychotic medications (e.g., chlorpromazine, thioridazine), antibiotics (e.g., gatifloxacin, moxifloxacin), or any other class of medications known to prolong the QTc interval. 6) Persistent elevation of liver function enzymes indicating active liver disease (elevated t. bilirubin > 1.5 mg/dl, or elevation to three-time normal range of liver enzymes, SGOT, SGPT, or g-GTP). 7) Any medication that is effective for alcohol dependence such as disulfiram, naltrexone, acamprosate, or topiramate. Carbamazepine for potential clinically significant drug-drug interaction. Other exclusion criteria include pregnancy, women who are breastfeeding, inability or unwillingness to use contraceptive methods, and inability to read or understand study forms and agrees to informed consent, or based on the judgment of the investigative team that the study may not be in the best interest of the subject either due to additional safety concerns or other factors that may interfere with study participations.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Paliperidone Palmitate Injection (INVEGA® SUSTENNA™) treated group will have a statistically significant advantage on improvement in manic symptoms. | 5 weeks
  This research can increase knowledge about the utility of paliperidone for improving symptoms of bipolar disorder and cravings of alcohol. If proven effective in reducing these symptoms, paliperidone could be a good and safe treatment option for dual diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ihsan Salloum, MD MPH, Principal Investigator — University of Miami